CLINICAL TRIAL: NCT02167542
Title: Positive Pressure During Bronchoscopy: Noninvasive Positive Pressure Ventilation vs Continuous Positive Airway Pressure Valve
Brief Title: Positive Pressure During Bronchoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Sao Joao (Other)
Responsible Party: Principal Investigator, Miguel R. Goncalves, PhD, Hospital Sao Joao
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BroncoNIVCPAP
Record Dates: First submitted 2011-09-15; First posted 2014-06-19 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Acute Respiratory Failure With Hypoxia
Keywords: Severe hypoxemic respiratory failure; Fiberoptic bronchoscopy; Noninvasive possitive pressure ventilation; Continuous positive airway pressure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NPPV group (Experimental): Patients assigned to noninvasive positive pressure ventilation (NPPV) are connected to the ventilator through a face mask (VBM Endoscopy Mask) that is secured to the patient's face by the investigator.
  Interventions: Device: Noninvasive Positive Pressure Ventilation
- CPAP valve group (Active Comparator): Patients assigned to CPAP valve (Boussignac valve, Vygon, Inc) are connected to this device through a standard face mask that is secured to the patient's face with elastic straps.
  Interventions: Device: CPAP valve (Boussignac)

INTERVENTIONS:
Device: Noninvasive Positive Pressure Ventilation — Patients assigned to NPPV were connected to the ventilator through a face mask (VBM Endoscopy Mask) that was secured to the patient's face by the investigator. Only one type of mechanical ventilator will be used (Vision, Philips Respironics). Ventilator parameters and supplemental oxygen will be titrated by the investigator to achieve SpO2>92%. Ventilatory support via face mask will be maintained with the same pressures for at least 30min after FOB, and then will be replaced by the FIO2 mask's if needed.
  Arms: NPPV group
Device: CPAP valve (Boussignac) — Patients assigned to CPAP Boussignac valve are connected to this device through a face mask that is secured to the patient's face with elastic straps. This kind of CPAP allows the delivery of pressure by constant-flow oxygen insufflation. Four funnel-shaped microchannels are included in the wall of this device and connected to an external opening connected to the oxygen source. These microchannels generate high-velocity microjets, which in turn generate the pressure resulting from the air entrainment mechanism thus created.
  Oxygen flow will be titrated by the investigator to ensure SpO2>92%.
  Arms: CPAP valve group

SUMMARY:
It has been demonstrated the application of noninvasive positive pressure ventilation (NPPV) to assist spontaneous breathing through a face mask during fiberoptic bronchoscopy (FOB) with bronchoalveolar lavage (BAL) in severely hypoxemic, nonintubated patients. With NPPV, FOB was well-tolerated, significantly improved the PaO2/FiO2 ratio, and successfully avoided the need for endotracheal intubation. Two randomized studies have provided supporting evidence that the application of NPPV or CPAP via a face mask was superior to oxygen supplementation alone during FOB.

For this reason patients who require FOB and are hypoxemic and/or mild hypercapnic (TcCO2 < 60mmHg) will be compared in a randomized study by comparing NPPV vs CPAP Boussignac (Vygon) delivered through a face mask.

DETAILED DESCRIPTION:
Since its introduction in the late 1960s, fiberoptic bronchoscopy (FOB) has been increasingly used for diagnostic and therapeutic purposes. Because arterial oxygen tension (PaO2) usually decreases by 10 to 20 mm Hg after uncomplicated bronchoscopy, severe hypoxemia in nonintubated patients is an accepted contraindication to bronchoscopy. The American Thoracic Society recommends avoiding bronchoalveolar lavage (BAL) in spontaneously breathing patients with hypercapnia or hypoxemia that cannot be corrected to at least a PaO2 of 75 mm Hg or to oxygen saturation greater than 90% with supplemental oxygen (1). In these high-risk patients, the options are to intubate and to apply mechanical ventilation (MV) to ensure adequate gas exchange during FOB or to avoid FOB and to institute empirical treatment.

This limitation has prompted the development of techniques of respiratory support to make the FOB procedure safer for hypoxemic or critically ill patients, without using invasive ventilation.

It has been demonstrated the application of noninvasive positive pressure ventilation (NPPV) to assist spontaneous breathing through a face mask during FOB with BAL in severely hypoxemic, nonintubated patients (2). FOB was well-tolerated, significantly improved the PaO2/FiO2 ratio, and successfully avoided the need for endotracheal intubation. Two randomized studies have provided supporting evidence that the application of NPPV or CPAP via a face mask was superior to oxygen supplementation alone during FOB (3,4).

For this reason patients who require FOB and are hypoxemic and/or mild hypercapnic (TcCO2 < 60mmHg) will be compared in a randomized study by comparing NPPV vs CPAP Boussignac (Vygon) delivered through a face mask.

Methods Adult patients will be recuited in Bronchology Department and Intensive Care Units of the Hospital S. João, EPE. Only when inclusion criteria and a written informed consent of participation have been obtained from the patient, they will enter this study.

Before undergoing bronchoscopy all patients will be evaluate by SpO2, TCCO2, arterial blood pressure (ABP), heart rate (HR), respiratory rate (RR) and ECG. Patients with SpO2<92%, oxygen supplementation will be provided to achieve SpO2>92%. At this stage all patients will be randomly assigned to receive NPPV or CPAP Boussignac through a face mask during bronchoscopy. During the procedure, patients will be continuous monitored with ECG, ABP, HR, RR, SpO2 and TCCO2. These clinical parameters will be recorded at the following times: 1 - at evaluation; 2 - before the beginning of FOB; 3 - during FOB; 4 - at the end of FOB; 5 - 5, 15, 30, 60 min after FOB.

ELIGIBILITY:
Inclusion Criteria:

* need for FOB;
* hypoxemia, defined by pulse oximetry (SpO2) >92% under oxygen supplementation;
* mild hypercapnia, defined by transcutaneous CO2 (PaCO2) <60mmHg;
* already under domiciliary NPPV.

Exclusion Criteria:

* emergent intubation;
* recent (less than 1 wk) acute myocardial infarction;
* ph bellow 7.30;
* PaCo2 > 60mmHg;
* systolic blood pressure < 80mmHg;
* encephalopathy or coma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-02; Primary Completion 2010-09 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change in arterial parcial oxygen pressure / Inspired oxygen fraction ratio (PaO2/FiO2) | Before and 5 min after the exam (FOB)

SECONDARY OUTCOMES:
Electrocardiogram | up to 60 min after FOB
Heart Rate | up to 60 min after FOB
Respiratory Rate | up to 60 min after FOB
Peripheal oxygen saturation | up to 60 min after FOB

CONTACTS AND LOCATIONS:
Overall Officials: Miguel R Gonçalves, Ph.D, Principal Investigator — Lung Function and Ventilation Unit, Pulmonology Department, University Hospital São João; Tiago F Pinto, MSc, Principal Investigator — Lung Function and Ventilation Unit, Pulmonology Department, University Hospital São João
Locations (1):
- Broncology Unit, Pulmonology Department, University Hospital São João, Porto, Porto District, Portugal

REFERENCES:
- [Background] Antonelli M, Conti G, Rocco M, Arcangeli A, Cavaliere F, Proietti R, Meduri GU. Noninvasive positive-pressure ventilation vs. conventional oxygen supplementation in hypoxemic patients undergoing diagnostic bronchoscopy. Chest. 2002 Apr;121(4):1149-54. doi: 10.1378/chest.121.4.1149. PMID 11948045